CLINICAL TRIAL: NCT00868595
Title: A Phase I, Non-randomized, Multiple Dose, Dose Escalation Study of the Safety, PK, PD and Efficacy of Therapeutic Vaccine, BP-GMAX-CD1, Plus Activating Agent, AP1903, in Patients With Castrate Resistant Prostate Cancer
Brief Title: MTD Study of Vaccine BP-GMAX-CD1 Plus AP1903 to Treat Castrate Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bellicum Pharmaceuticals (Industry)
Collaborators: M.D. Anderson Cancer Center (Other); The University of Texas Health Science Center, Houston (Other); Memorial Hermann Hospital (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP-PC-001
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Castrate Resistant Prostate Cancer (CRPC)
MeSH Terms: interventions — AP 1903 reagent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): Cohort 1: BPX-101, 4 x 10*6 cells administered every other week for 6 cycles Cohort 2: BPX-101, 12.5 x 10*6 cells administered every other week for 6 cycles Cohort 3: BPX-101, 25 x 10*6 cells administered every other week for 6 cycles Cohort 4: BPX-101, 25 x 10*6 cells administered every 4 weeks for 3 cycles
  At 24 hours after each vaccination, a single dose of the activating agent, AP1903 for Injection, will be administered at a fixed dose of 0.4 mg/kg via intravenous (IV) infusion over 2 hours.
  Interventions: Biological: BPX-101; Drug: AP1903

INTERVENTIONS:
Biological: BPX-101 — Vaccine
  Other Names: N/Ap
Drug: AP1903 — Activating agent, infusion
  Other Names: N/Ap

SUMMARY:
This is a Phase I, non-randomized, multiple-dose, 3+3 dose-escalation study of the safety, pharmacokinetics, biomarkers, preliminary efficacy and patient-reported outcomes of therapeutic vaccine, BPX-101 (formerly BP-GMAX-CD1), plus activating agent, AP1903, in patients with castrate resistant prostate cancer.

DETAILED DESCRIPTION:
Patients will be screened within 6 weeks prior to Week 1. A total of 3 cohorts, consisting of 3 to 6 patients each, are planned to receive five to eight intradermal (ID) injections totaling 1 mL up to 1.6mL of BPX-101 at 3 doses levels for an initial 6 doses.

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥ 18 years of age
2. Histological diagnosis of adenocarcinoma of the prostate
3. Documented evidence of distant metastasis of disease
4. No more than 1 prior chemotherapeutic, biologic or combination treatment regimen (including vitamin D analogues) for CRPC. If previously treated, patients must be recovered from all toxicities prior to entry into the study.
5. Patients must have current or historical evidence of disease progression concomitant with surgical (orchiectomy) or medical castration (LHRH analogue); anti-androgen withdrawal (4 weeks for flutamide and 6 weeks for nilutamide or bicalutamide) is necessary only for patients on antiandrogens and a duration of response to antiandrogens > 3months;
6. Testosterone < 50 ng/dL achieved via medical or surgical castration. Patients receiving medical castration therapy must continue such therapy throughout the study.
7. Adequate hematologic, renal and liver function:
8. Negative serology tests for human immunodeficiency virus (HIV-1 and 2), human T-cell lymphotropic virus (HTLV-1), hepatitis B surface antigen (HBsAg) and hepatitis C (HCV)
9. Karnofsky Performance Score (KPS) ≥ 70%
10. Life expectancy > 6 months
11. Written informed consent obtained prior to the initiation of study procedures

Exclusion Criteria:

1. The presence of brain metastases, pleural effusions or ascites
2. Pathologic long-bone fractures, imminent pathologic long-bone fracture (cortical erosion on radiography > 50%), or spinal cord compression
3. A history of stage III or greater cancer, excluding prostate cancer. Basal or squamous cell skin cancers must have been adequately treated and the patient must be disease-free at the time of registration. Patients with a history of stage I or II other cancers must have been adequately treated and been disease-free for 3 years at the time of registration.
4. More than 1 prior chemotherapy, biologic or combination treatment regimen (including vitamin D analogues) for CRPC
5. Any treatment with radiopharmaceuticals, e.g. Strontium-89 and Samarium-153
6. Ketoconazole or antiandrogens (flutamide, nilutamide, bicalutamide) within 2 weeks prior to registration. Patients who demonstrate an anti-androgen withdrawal response, defined as a > 25% drop in PSA within 4 weeks (flutamide) or 6 weeks (nilutamide, bicalutamide) of stopping a non-steroidal anti-androgen, are not eligible until the PSA rises above the nadir observed after anti-androgen withdrawal.
7. Initiation of bisphosphonate therapy within 28 days prior to registration. Patients taking bisphosphonates should not have their dosing regimen altered unless medically warranted.
8. A requirement for systemic steroid or other immunosuppressive therapy for any reason.
9. Treatment with any of the following medications or interventions < 28 days prior to Screening
10. Treatment with any investigational vaccine within 2 years prior to Screening, or treatment with any other investigational product within 28 days prior to Screening
11. Any antibiotic therapy or infection within 1 week prior to Screening, including unexplained fever (temperature ≥ 100.5F or 38.1C)
12. History of autoimmune disease
13. Serious ongoing chronic or acute illness
14. Any medical intervention or other condition which, in the opinion of the Principal Investigator and/or the Bellicum Medical Monitor, could compromise adherence with study requirements

Other Criteria Apply however are not listed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-04; Primary Completion 2011-07 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of BPX-101 and AP1903 | 1 Year
  To determine the maximum tolerated dose (MTD) of BPX-101 and AP1903 when administered 24 hours apart
Safety and tolerability of BPX-101 and AP1903 | 1 Year
  To determine other measures of safety and tolerability of BPX-101 and AP1903 when administered 24 hours apart to patients with castrate resistant prostate cancer (CRPC).

SECONDARY OUTCOMES:
Pharmacokinetics of AP1903 | 1 Year
  To determine the pharmacokinetics of AP1903 when administered 24 hours after BPX-101
Immune responses and their association with clinical outcome | 2 Years
  To assess immune responses and their association with clinical outcome as measured by changes in levels of interferon gamma (IFN)-producing T cells, the cytotoxic T lymphocyte (CTL) response, cytokines (IFN, IL-4, IL-10), activation markers, and other markers
PSA response and PSA dynamics | 1 Year
  To assess PSA response and PSA dynamics (change in velocity, doubling time)
Number of circulating tumor cells (CTC) | 1 Year
  To assess reduction in the number of circulating tumor cells (CTC)
Cancer-related pain | 1 Year
  To assess cancer-related pain
Pain medication usage | 1 Year
  To assess pain medication usage
Preliminary efficacy of BPX-101 at the maximum tolerated dose (MTD) | 2 Years
  To determine preliminary efficacy of BPX-101 at the maximum tolerated dose (MTD), based on tumor assessments using computed tomography (CT) or magnetic resonance imaging (MRI) and radionuclide bone scans

CONTACTS AND LOCATIONS:
Overall Officials: Guru Sonpavde, MD, Principal Investigator — University of Texas Health Science Center Houston - CCTS
Locations (1):
- University of Texas Health Science Center Houston, CRU, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Bellicum Pharmaceuticals Home Page — http://www.bellicum.com/